CLINICAL TRIAL: NCT02020161
Title: Clinical Guidelines for APL Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETHEMA LPA2012
Record Dates: First submitted 2013-11-26; First posted 2013-12-24 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: APL
MeSH Terms: interventions — Tretinoin; Idarubicin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATRA-Idarubicin (Experimental)
  Interventions: Drug: Atra; Drug: Idarubicin; Drug: methotrexate

INTERVENTIONS:
Drug: Atra
Drug: Idarubicin
Drug: methotrexate

SUMMARY:
Therapeutic guidelines for treatment of patients with de novo APL to be used by every institution that wants to follow them. All patients who are reported may be retrospectively analyzed

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of acute promyelocytic leukemia

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence within 1 year of treatment | 3 years
  Induction therapy with simultaneous ATRA (45 mg/m2 day until CR) and idarubicin (12 mg/m2 day on days 2, 4, 6 and 8 or 12 mg/m2 day on days 2, 4 and 6 in patients older than or equal to 60 years).
  Three monthly consolidation courses with ATRA Maintenance therapy with ATRA (45 mg/m2/d, days 1-15 every 3 months), and low dose chemotherapy with methotrexate (15 mg/m2/d, weekly) and 6-mercaptopurine (50 mg/m2/d) for two years.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Fe, Valencia, Spain